CLINICAL TRIAL: NCT03664687
Title: A Randomised, Multicentre, Pragmatic Trial Comparing a Single-Dose vs. Twice Yearly Zoledronate in Patients With Early Stage Breast Cancer (REaCT-ZOL)
Brief Title: Comparing a Single-Dose vs. Twice Yearly Zoledronate in Patients With Early Stage Breast Cancer (REaCT-ZOL)
Acronym: REaCT-ZOL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OTT 18-01
Record Dates: First submitted 2018-09-06; First posted 2018-09-10 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Early-stage Breast Cancer
Keywords: Adjuvant Zoledronate
MeSH Terms: conditions — Breast Neoplasms | interventions — Zoledronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Zoledronate one dose (4 mg) (Active Comparator): One 4 mg dose of Zoledronate
  Interventions: Drug: Zoledronate
- Zoledronate 4 mg every 6 months x 3 years (Active Comparator): One 4 mg dose of Zoledronate given every 6 months for 3 years
  Interventions: Drug: Zoledronate

INTERVENTIONS:
Drug: Zoledronate — Administered intravenously (IV)
  Other Names: Zoledronic acid

SUMMARY:
REaCT ZOL will compare one 4 mg dose of Zoledronate vs. one 4 mg dose of Zoledronate given every 6 months for 3 years.

DETAILED DESCRIPTION:
Breast cancer patients are at an increased risk of recurrence in bone and bone density loss (osteopenia/osteoporosis) and consequently fragility fractures due to: age, systemic therapy with aromatase inhibitors, and premature induction of menopause by chemotherapy or ovarian ablation. Bone is the most common site of breast cancer recurrence. The use of bone modifying agents, such as Zoledronate may reduce the risk of bone metastases and fragility fractures. Despite the widespread use of adjuvant Zoledronate, it is not known what the optimal number of infusions is to reduce the risk of bone metastases and the risk of fragility fractures. Indeed, the recent CCO and ASCO Practice Guideline, 'Bottom line recommendations' specifically states, "More research is recommended comparing different bone-modifying agents, doses, dosing intervals, and durations." In the metastatic setting, for nearly 2 decades biphosphonates (i.e. Zoledronate) have been given to patients every 3-4 weeks. This dosing interval was selected based on convenience of co-administration with standard anti-cancer agents and not on the long biological effect of these agents on osteoclasts, the cells responsible for excess bone breakdown. Furthermore, in the bone density preservation setting, despite the usual administration of Zoledronate once a year a single dose of Zoledronate was associated with a sustained increase in bone mineral density 5 years later. A recent systematic review in the adjuvant setting, showed that BTA at any particular dose or route of administration showed superiority over the other. In other words, the lowest dose appears to be just as good as the highest dose. This study will compare the single dose of Zoledronate to Zoledronate given every 6 months for 3 years. The primary outcome for this study will be feasibility of conducting this trial. The secondary outcome will assess bone-metastasis risk, fragility rates, quality of life, and cost-effectiveness.

In this study it is hypothesized that a single dose of Zoledronate will be non-inferior to every 6 months in terms of bone-metastasis free survival, time to first bone metastasis and fragility fractures. It is also hypothesized that a single dose of Zoledronate will have less toxicities associated with Zoledronate compared to every 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Commencing zoledronate within 3 months of starting neoadjuvant or adjuvant endocrine therapy or within 3 months of completion of neoadjuvant or adjuvant chemotherapy for early stage breast cancer
* Patients receiving any intravenous or oral biphosphonates, or subcutaneous denosumab for the treatment of osteoporosis must discontinue treatment prior to baseline evaluation
* ECOG performance status equal or less than 2 and life expectancy of more than 12 months
* Serum creatinine greater than 30 ml/min and corrected serum calcium equal or greater than 2 mmol/l within 4 weeks before first zoledronate infusion
* Age equal or greater than 18 years
* Able to provide written consent

Exclusion Criteria:

* Metastatic disease
* History of osteonecrosis of the jaw
* Known hypersensitivity to trial drug or hypersensitivity to any other component of the trial drug (e.g. fructose)
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the trial protocol
* Pregnancy or risk of pregnancy (this includes participants that are not willing to practice active contraception for the duration of the study)* *Women/men of child bearing potential must have agreed to use two effective contraceptive methods while on study. A women is considered to be of 'childbearing potential' if she has had menses at any time in the preceding 12 consecutive months. In addition to routine contraceptive methods. 'effective contraception' also includes heterosexual celibacy and surgery intended to prevent pregnancy (or with a side-effect of pregnancy prevention) defined as complete hysterectomy, bilateral oophorectomy or bilateral tubal ligation, or vasectomy/vasectomized partner. However, if at any point a previously celibate participant chooses to become heterosexually active during the period for use of contraceptive measures outlined in the protocol, she is responsible for beginning contraceptive measures. Examples of effective methods of contraception: Male condom plus spermicide; Cap plus spermicide; Diaphragm plus spermicide; intrauterine device (Copper T, Progesterone T; Levonorgestrel-releasing intrauterine system (i.e. Mirena); hormonal methods (implants, hormonal shot or injection, combined pill, minipill, patch).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2018-10-31 (Actual); Primary Completion 2020-04-02 (Actual); Study Completion 2025-03-28 (Actual)

PRIMARY OUTCOMES:
Multiple Site Activation | 12 months
  Evaluating the feasibility of multiple site activation. Measured by the number of sites activated, as well as how long it takes to get the sites activated once the first site becomes active for accrual.
Time to Activate Six Sites | 12 months
  Evaluating the amount of time it takes to get six sites activated for participant accrual.
Medical Oncologist Active Participation | Through to end of accrual, average 2 years
  Evaluating the number of medical oncologists at each study site who actively participate in the trial. Active participation includes approaching eligible patients for the study, as well as following up with patients who are taking part in the study.
Patient Enrollment | 9 months
  Evaluating the number of patients enrolled across all of the active sites within 9 months of the sixth site being activated. Number of patients enrolled across all of the active sites.

SECONDARY OUTCOMES:
Bone-Metastasis-Free Survival | Through to end of study, average of 3 years
  Evaluate bone-metastasis-free Survival (Bone-DFS) defined as the time to first occurrence of bone metastasis (symptomatic or asymptomatic) or death from any cause.
Time to first bone metastasis | Through to end of study, average of 3 years
  Evaluate the time to first bone metastasis (symptomatic or asymptomatic, excluding deaths). The time-to-disease will start from the randomization data and ends at occurrence of the event.
Fragility fractures rates | Through to end of study, average of 3 years
  Evaluate fragility fracture rates. Fragility fractures rates; defined as fractures which result from a fall from a standing height or less, or that present in the absence of trauma (most common fragility fractures occur at the hip, wrist, spine, humerus or pelvis).
Direct Estimation of Health Utility Values | Through to end of study, average of 3 years
  To evaluate patient quality of life using the EQ-5D-5L questionnaire, undertaken at the first Zoledronate treatment and either every year (Arm A) or every 6 months (Arm B) for 3 years. The EuroQol 5 Dimension 5 Level (EQ-5D-5L) questionnaire consists of two sections; the descriptive system and the visual analogue scale. The descriptive system comprises 5 dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) and has 5 levels associated with it (no problems, slight problems, moderate problems, severe problems and extreme problems). The scale range of 1-5 is used for the 5 dimensions where 1 is the best outcome and 5 is the worst outcome. The Visual Analogue scale records the respondent's self-rated health on a vertical, visual scale with endpoints labelled 'the best health you can imagine' at the top and 'the worst health you can imagine' at the bottom. This ranges 0-100 with 0 being the worst outcome and 100 being the best outcome.
Incremental Cost-Effectiveness Ratio | Through to study completion, an average of 3 years
  A statistic used in cost-effectiveness analysis to summarise the cost-effectiveness of a health care intervention. It is defined by the difference in cost between two possible interventions, divided by the difference in their effect.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Clemons, MD, Principal Investigator — Ottawa Hospital Research Institute
Locations (6):
- Canada (6):
  - William Osler Health System, Brampton Civic Hospital, Brampton, Ontario
  - Juravinski Cancer Centre, Hamilton, Ontario
  - Kingston Health Sciences Centre, Kingston, Ontario
  - Markham Stouffville Hospital, Markham, Ontario
  - Southlake Regional Health Centre, Newmarket, Ontario
  - Ottawa Hospital Research Institute, Ottawa, Ontario

REFERENCES:
- [Background] Awan A, Ng T, Conter H, Raskin W, Stober C, Simos D, Pond G, Dhesy-Thind S, Mates M, Kumar V, Fergusson D, Hutton B, Saunders D, Vandermeer L, Clemons M; REaCT Investigators. Feasibility outcomes of a randomised, multicentre, pilot trial comparing standard 6-monthly dosing of adjuvant zoledronate with a single one-time dose in patients with early stage breast cancer. J Bone Oncol. 2020 Dec 13;26:100343. doi: 10.1016/j.jbo.2020.100343. eCollection 2021 Feb. PMID 33425673
- [Background] McGee S, Alzahrani M, Vandermeer L, Cole K, Larocque G, Awan A, Hutton B, Pond G, Saunders D, Clemons M. Adjuvant bisphosphonate use in patients with early stage breast cancer: a physician survey. Breast Cancer Res Treat. 2021 Jun;187(2):477-486. doi: 10.1007/s10549-021-06147-1. Epub 2021 Mar 23. PMID 33755864
- [Background] McGee S, AlZahrani M, Stober C, Ng TL, Cole K, Larocque G, Awan A, Sehdev S, Hilton J, Vandermeer L, Hutton B, Pond G, Saunders D, Clemons M. Adjuvant bisphosphonate use in patients with early stage breast cancer: Patient perspectives on treatment acceptability and potential de-escalation. J Bone Oncol. 2021 Feb 19;27:100351. doi: 10.1016/j.jbo.2021.100351. eCollection 2021 Apr. PMID 33680749
- See also: The Rethinking Clinical Trials (REaCT) website — https://react.ohri.ca/